CLINICAL TRIAL: NCT05170490
Title: Long Term Follow up of Chronic Hepatitis C Patients Treated With Direct Acting Antivirals After Sustained Virological Response
Brief Title: Long Term Follow up of Chronic HCV Patients Receiving DAAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amira Maher, Lecturer, Sohag University
Other Study IDs: DAAS in HCV patients
Record Dates: First submitted 2021-12-24; First posted 2021-12-28 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Chronic Hepatitis c
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Follow up of Chronic hepatitis C Patients with moderate to severe fibrosis and cirrhosis treated with Direct Acting Antivirals after Sustained Virological Response for 4-5 years to detect changes in hepatic fibrosis and liver functions.

DETAILED DESCRIPTION:
Treatment of chronic hepatitis C is evolving rapidly. Three classes of direct-acting antiviral agents, including inhibitors of the HCV NS3/4A protease, NS5B polymerase, and NS5A have been approved for the treatment of patients with chronic hepatitis C, both in combination with pegylated Interferon (Peg-IFN) / ribavirin (RBV) and, recently, in interferon-free combination.

The objective of chronic hepatitis C treatment is to achieve SVR which is defined as the absence of viral replication at 12 or 24 weeks after treatment completion. SVR reduces morbidity and mortality and is equivalent in most cases to cure the HCV infection. Studies have demonstrated that SVR is associated with histological improvement, assessed by liver biopsy, and with the prevention of complications, such as the development of liver cirrhosis and HCC.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HCV patients with moderate to severe hepatic fibrosis (F2: F4) or cirrhosis who received direct-acting antivirals and achieved SVR.

Exclusion Criteria:

* Other liver diseases as Chronic hepatitis B and autoimmune liver disease. HIV co-infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with chronic hepatitis C who received direct-acting antiviral drugs and scheived SVR
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
changes in hepatic fibrosis | 4 years after end of treatment
  Shear wave elastography

SECONDARY OUTCOMES:
change in serum albumin level | 4 years after end of treatment
  change in liver function
change in prothrombin level | 4 years after end of treatment
  change in liver function
change in bilirubin level | 4 years after end of treatment
  change in liver function

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No